CLINICAL TRIAL: NCT05024305
Title: A Multi-center, Phase I, Open Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Efficacy of TWP-102 in Patients With Advanced Malignancies.
Brief Title: Safety, Tolerability, PK, PD, Immunogenicity and Efficacy of TWP-102 in Patients With Advanced Malignancies.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong TheraWisdom Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TWP-102-11
Record Dates: First submitted 2021-08-22; First posted 2021-08-27 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-08

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Four dose levels of TWP-102 injection will be tested by BOIN study design.
  Interventions: Drug: TWP-102 injection
- Dose Expansion Cohort (Experimental): Once the effective doses have been determined, two expansion cohorts will be opened to evaluate the efficacy and safety in one or two tumors.
  Interventions: Drug: TWP-102 injection

INTERVENTIONS:
Drug: TWP-102 injection — IV infusion

SUMMARY:
This is a multi-center, phase I, open clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity and efficacy of TWP-102 injection in patients with advanced malignancies. This study consists of two parts, including a dose escalation study and a dose expansion study. The criteria for dose escalation will be based on the Bayesian optimal interval (BOIN) design with sequentially enrolled cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced malignancies that failed, or not suitable for standard treatments;
* At least 1 measurable lesion.
* ECOG score 0 or 1;
* Life expectancy of ≥ 3 months;

Exclusion Criteria:

* Known hypersensitivity to any ingredient of TWP-102;
* Receiving any anti-cancer drugs within 4 weeks;
* History of serious systemic diseases;
* History of serious autoimmune diseases;
* Persistent toxicity of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade > 1 severity that is related to prior anti-cancer therapy. (except alopecia)
* Pregnancy or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events/serious adverse event related with TWP-102 injection | From enrollment until 90 days after the last dose
Dose-limiting toxicity (DLT) | From the first dose of study drug up to 3 weeks

SECONDARY OUTCOMES:
Maximum measured plasma concentration (Cmax) of TWP-102 injection. | From first dose until 90 days after the last dose
Time to maximum plasma concentration (Tmax) of TWP-102 injection. | From first dose until 90 days after the last dose
Half-life (T1/2) of TWP-102 injection. | From first dose until 90 days after the last dose
Immunogenicity profile of TWP-102 injection. | From first dose until 90 days after the last dose
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies and neutralizing antibodies.
Objective Response Rate (ORR) | From first dose to disease progression or end of study, an average of 2 years
Duration of Response (DOR) | From first dose to disease progression or end of study, an average of 2 years
Disease control rate (DCR) | From first dose to disease progression or end of study, an average of 2 years
Progression free survival (PFS) | From first dose to disease progression or end of study, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China